CLINICAL TRIAL: NCT06435182
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Safety and Efficacy of OT202 Eye Drops in the Treatment of Moderate to Severe Dry Eye
Brief Title: Study of OT202 in Treating Moderate to Severe Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocumension Therapeutics (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ocumension Therapeutics (Suzhou) Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OT202-02-01
Record Dates: First submitted 2024-05-20; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Dry Eye
Keywords: Moderate dry eye; Severe dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Parallel assignment: 0.5% OT202 eye drop group；1% OT202 eye drop group；OT202 solvent eye drop group with a 1:1:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OT202 conc.0.5% group (Experimental): Administered three times daily (morning, afternoon, and evening), with 1-2 drops each time, instilled into the conjunctival sac.
  Interventions: Drug: OT202 conc 0.5%
- OT202 conc. 0.1% group (Experimental): Administered three times daily (morning, afternoon, and evening), with 1-2 drops each time, instilled into the conjunctival sac.
  Interventions: Drug: OT202 conc 0.1%
- Placebo group (Experimental): Administered three times daily (morning, afternoon, and evening), with 1-2 drops each time, instilled into the conjunctival sac.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OT202 conc 0.5% — Apply 1-2 drops of OT202 0.5% solution into the conjunctival sac. three times daily
  Other Names: Investigational product
  Arms: OT202 conc.0.5% group
Drug: OT202 conc 0.1% — Apply 1-2 drops of OT202 0.1% solution into the conjunctival sac. three times daily
  Other Names: Investigational product
  Arms: OT202 conc. 0.1% group
Drug: Placebo — Apply 1-2 drops of placebo solution into the conjunctival sac. three times daily
  Arms: Placebo group

SUMMARY:
This is a phase II study to explore the optimal dosage of OT202 in treating dry eye.

DETAILED DESCRIPTION:
Subjects successfully enrolled will enter a 2-week induction period of OT202 solvent eye drops, treated with OT202 three times daily (morning, afternoon, and evening), with 1-2 drops each time. On the day of the baseline visit (Visit 2), subjects will be assessed again to meet the inclusion and exclusion criteria. Subjects remain in the study are then randomized with a 1:1:1 ratio to 3 groups, the 0.5% OT202 eye drop group, 1% OT202 eye drop group, or OT202 solvent eye drop group, for an 8-week treatment period. Safety visits will be conducted 2 weeks after completion of the respective treatment.

ELIGIBILITY:
---Inclusion Criteria ---

1. 18 to 75 years of age (inclusive) at the time of signing the ICF, either sex or ethnic group.
2. With history of dry eye for at least 6 months prior to screening, and history of use or willingness to use eye drops for the treatment of dry eye within 6 months prior to screening

   .
3. Binocular BCVA ≥ 0.25 decimals (standard logarithmic visual acuity chart) at Screening and Baseline.
4. At least one eye (the same eye) meets all the following criteria at screening and baseline:

   * TCSS ≥ 2 points
   * Eye dryness score (EDS) ≥ 40 points in VAS
   * Conjunctival hyperemia score ≥ 1 point
   * TFBUT ≤ 5 seconds
   * 1 mm/5 min ≤ Schirmer I test (without surface anesthesia) ≤ 10 mm/5 min
5. Must be able to understand and sign the ICF approved by Independent Ethics Committee (EC).
6. Willing and able to conduct protocol-required study visits, follow study guidelines, and take study drug as instructed.

---Exclusion Criteria ---

1. With contraindication or hypersensitivity to the study drug (OT202 and excipients) or diagnostic reagents (fluorescein sodium, lissamine green, etc.).
2. During the screening period and baseline period, any eye with ocular active inflammation or structural abnormalities that may affect the trial assessment, including but not limited to trichiasis, blepharospasm, blepharitis, meibomitis, severe meibomian gland dysfunction, bulbar conjunctival laxity, keratitis, recurrent corneal erosion, allergic conjunctivitis, iritis, anterior chamber inflammation, known retinal detachment, diabetic retinopathy, or history of any progressive retinal disease.
3. With history of possible or confirmed ocular infection (bacterial, viral, or fungal) or ocular herpes (simple or zoster) in either eye, as determined by the patient's medical history and/or at the screening and baseline examinations.
4. Those with intraocular pressure (non-contact tonometry) greater than 21 mmHg or less than 8 mmHg or diagnosed with glaucoma at screening and baseline, or those with ocular hypertension who underwent intraocular pressure reduction therapy, and those with a history or suspicion of glaucoma.
5. Those with any systemic disease expected to potentially affect the study results. It include but is not limited to Sjögren syndrome, Stevens-Johnson syndrome, rheumatoid arthritis, graft versus host disease, systemic lupus erythematosus, scleroderma, sarcoidosis, herpes, acne, rosacea, etc.
6. Those who cannot stop using any ocular medication or treatment during the clinical trial.
7. Those with recent clinically relevant history (e.g., hepatic, renal impairment) within 6 months prior to screening or current severe, unstable, or uncontrolled cardiovascular, pulmonary, hepatic, renal, autoimmune, and other relevant systemic diseases (e.g., severe chronic obstructive pulmonary disease, arrhythmia, significant heart failure, uncontrolled hypertension, type 2 diabetes mellitus), as assessed by the investigator.
8. Those on a chronic, systemic medication regimen used for less than 1 month at screening and baseline or with dose changed within 1 month (including initiation of new medication and discontinuation).
9. Those who have used any prohibited medications (topical ocular, systemic, and/or injectable medications) during the specified period prior to screening. These medications are also prohibited during the study. However, if a subject has a prohibited medication at screening, it needs to be stopped and washed out according to the washout period specified below, which can be included in the wash-out period. The minimum reasonable washout period for prohibited medications is as follows:

   * Systemic and local immunosuppressant and immunotherapy (such as cyclosporine eye drops, tacrolimus eye drops, etc.): 60 days;
   * Corticosteroids (any route): 14 days;
   * Systemic or ocular topical mast cell stabilizers, antihistamines, antihistamines/mast cell stabilizer combination, vasoconstrictors, monoamine oxidase inhibitors: 7 days;
   * Other topical ophthalmic preparations (including artificial tears): 3 days;
   * Medications known to cause ocular dryness (e.g., anticholinergics, serotonin reuptake inhibitors, beta-blockers, diuretics, etc.): 14 days.

   Note:Non-periocular, low-potency, over-the-counter corticosteroid topical skin creams are allowed for use in the study (e.g., hydrocortisone butyrate cream/ointment).
10. Previous use of spleen tyrosine kinase (Syk) inhibitors or eye drop products targeting the same as anti-vascular endothelial growth factor (VEGF).
11. Those who wore corneal contact lenses within 7 days prior to screening or required them during the study.
12. Those who underwent meibomian gland massage or moist chamber therapy within 7 days prior to screening, or non-drug therapies for dry eye such as intense pulsed light therapy, thermal pulsation therapy, etc., within the previous 6 months before screening.
13. Those who previously underwent dry eye surgery such as tear duct embolization (current tear duct embolization status or punctal plug use in the past 6 months) or amniotic membrane transplantation.
14. Those who underwent ocular surface surgery (e.g., LASIK excimer laser in situ keratomileusis) within 12 months prior to screening or intraocular surgery within 6 months prior to screening in either eye, as determined by the subject's medical history and/or examination, or anticipated ocular surgery during the study.
15. Those who use other investigational products or devices within 3 months prior to screening or concurrently during the study.
16. Non-compliance with drug administration (< 80% or > 120%) during the introduction period.
17. Females of childbearing potential who are currently pregnant, or have a positive pregnancy test result, or plan to get pregnant during the study, or are currently breastfeeding, or do not agree to use appropriate contraception methods to avoid pregnancy during the study period up to 1 month after the last dose of study drug.
18. Males who do not agree to use one or more acceptable effective contraception methods during the study period up to 1 month after the last dose of study drug.
19. Any condition or situation that, in the opinion of the investigator, may pose a safety risk to the subject in the trial or may interfere with the conduct of the study, or the investigator believes that the subject may not be able to complete or comply with the requirements of the study (due to administrative reasons or otherwise).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Total Corneal Fluorescein Staining (TCSS) score | Day 56
  Compare the difference of changes in TCSS relative to baseline of three study groups on day 56.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) Score | DAY 28 & 56
  Compare the difference of changes in VAS scale relative to baseline of three study groups on day 28 & 56.
Ocular Surface Disease Index (OSDI) Score | Day 28 & 56
  Compare the DAY 28 & 56 OSDI scale results of the subjects with the baseline results.
Conjunctive Hyperemia | Day 28 & 56
  Compare the DAY 28 & 56 Conjunctive Hyperemia data of the subjects with the baseline data.
Corneal Staining | Day 28 & 56
  Compare the DAY 28 & 56 Corneal Staining data of the subjects with the baseline data.
A dry eye syndrome questionnaire - Symptom Assessment iN Dry Eye(SANDE) | Day 28 & 56
  Compare the DAY 28 & 56 SANDE scale results of the subjects with baseline .
Tear Film Breakup-time (TFBUT) | Day 28 & 56
  Compare the DAY 28 & 56 TFBUT scale results of the subjects with baseline .
Schirmer I Test | Day 28 & 56
  Compare the DAY 28 & 56 Schirmer I Test scale results of the subjects with baseline .

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, Principal Investigator — Eye Hospital, WMU; Jialu Xia, Study Director — Sponsor GmbH
Locations (10):
- China (10):
  - The Third Xiangya Hospital Of Central South University, Changsha
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Then Second People's Hospital of Yunnan Province, Kunming
  - Ning Bo Eye Hospital, Ningbo
  - Tianjin Eye Hospital, Tianjin
  - Tianjin Medical University Eye Hospital, Tianjin
  - Eye Hospital, WMU, Wenzhou
  - Renmin Hospital of Wuhan University, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an

IPD SHARING:
Plan to Share IPD: No